CLINICAL TRIAL: NCT05591248
Title: Virtual Reality Rehabilitation (VRR) on the Intensive Care Unit (ICU) for Critically Ill Patients: a Feasibility Study and Further Development of the "MotiVeeR UZeLf"-App
Brief Title: Virtual Reality Rehabilitation on the Intensive Care Unit for Critically Ill Patients
Acronym: VRR-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S66360
Record Dates: First submitted 2022-09-28; First posted 2022-10-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Critical Illness; Intensive Care Unit Acquired Weakness
Keywords: Virtual Reality; Rehabilitation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group Virtual Reality Rehabilitation (Experimental): All included patients will receive 3 - 9 sessions (3x/w) of VR rehabilitation during their stay at the intensive care unit. The games will stimulate them to move the arm(s). How long they play the game(s) is not decided in advance (patient-therapist-decision at the time of playing).
  Interventions: Device: VRR

INTERVENTIONS:
Device: VRR — Eligible patients meeting the inclusion criteria and signed a consent, will have 3x/week the guided rehabilitation session with the VR-tool (with a maximum of 9 VRR-sessions).

SUMMARY:
Feasibility study of the use of an interactive Virtual Reality device in rehabilitation of critically ill patients on the Intensive Care Unit. Patients will use the upper limb muscles and memory playing the 2 games in our "MotiVeeR UZeLf"-app. This will be the case 3x/week as part of the conventional rehabilitation program.

DETAILED DESCRIPTION:
Virtual Reality (VR) is the simulation of a real environment generated by a computer software and experienced by the user through glasses that are slid over the head. VR is already known for its use in the entertainment and technology industry, but there is a growing interest in the use of VR for medical purposes. Also in the field of rehabilitation, virtual reality rehabilitation (VRR) has been studied in different patient populations, with beneficial effect.

For intensive care, VRR is a new but promising application domain. Patients in intensive care (IC) need specific medical care and rehabilitation. Critically ill patients who are in an intensive care for a long time (8 or more days) often show a severe muscle weakness caused by being critically ill in itself.

The importance and benefits of starting rehabilitation as soon as possible has been undeniably established in the literature. Early mobilization and exercises during the stay at IC prevents the occurrence of muscle weakness or reduces its onset, shortens the duration of the stay at IC and improves functionality.

In addition to the muscle problems, changes in the brain or impaired mental functioning can also occur in IC patients.

A rehabilitation program for ICU patients that stimulates memory and attention, combined with physical and functional training, could potentially be effective in improving mental performance and functional outcomes.

The investigators will record the time required for the setup, learning, use and cleaning of the advanced device, and note any problems that delay this process. Patients will be encouraged to report any type of problem (technical, medical, emotional) at any time (before/during/after the procedure). Any problem spontaneously reported by the patient will be registered. The study will cover the virtual world in a closed headset, completely blocking any other vision, while the patient will be encouraged/triggered to move the arms. The feasibility and safety of using such a closed VR headset on IC patients during rehabilitation exercises is being studied.

Many of the VR modules available today are focused on passive forms of VR, with the aim of relaxation. With this project, the investigators created an interactive ICU-specific VRR app, using a closed VR headset, to stimulate motivation for muscle and attention training in ICU patients through a game.

The exercise program will be gradually build up from low to medium training intensity. Only the therapist (and not the patient) can change the level of difficulty/intensity, so that a correct training intensity is guaranteed.

With this study the investigators want to test whether this form of support of exercise therapy is feasible and safe in Intensive Care. The investigators also want to test whether the patient and the physiotherapist / occupational therapist remain motivated with this VRR for exercise therapy, also for bedridden ICU patients with a long stay.

ELIGIBILITY:
Inclusion Criteria:

* Admission to surgical ICU >= 3 days, with a prognosis of ICU admission at least 2 more weeks
* Adult
* Alert and calm (RASS -1 to +1)
* Adequate (Standard 5 Questions; S5Q >= 4/5)
* Indication for rehabilitation therapy
* Able to lift (at least) 1 arm against gravity

Exclusion Criteria:

* Blind
* Schizophrenia, advanced dementia, dissociative disorder, serious claustrophobia
* Age < 18 years and/or mental age < 18 years
* Incapacity
* Pregnancy
* No understanding of Dutch or French or English
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety of VRR on ICU? (Adverse Events?) | Inclusion between 31/10/2022 and 31/10/2023. Screening for this particular outcome will happen during the 3-week-VR-training period for each patient.
  Screening for minor and major adverse events of VRR on ICU patients.
Feasibility (related to time) of VRR on ICU? | Inclusion between 31/10/2022 and 31/10/2023. Screening for this particular outcome will happen during the 3-week-VR-training period for each patient.
  Time needed for set-up, explication, use and cleaning of the device will be registrated (in minutes). Set-up or explication or cleaning taking longer than 15min will be labeled as 'not feasible'.
Feasibility (related to practicability) of VRR on ICU? | Inclusion between 31/10/2022 and 31/10/2023. Screening for this particular outcome will happen during the 3-week-VR-training period for each patient.
  Screening for technical/practical/logistical issues will happen through a self-made (and by protocol accepted) questionnaire. For every question there is a 5-point Likert Scale (1 meaning "not at all" and 5 meaning "very much") that needs to be answered.

SECONDARY OUTCOMES:
Patient's satisfaction of the use of VR as a tool for rehabilitation on ICU | Inclusion between 31/10/2022 and 31/10/2023. Screening for this particular outcome will happen during the 3-week-VR-training period for each patient + 1 month after ICU-discharge.
  Motivation, happiness, ... (through self-made questionnaire based on existing literature and approved by protocol). For every question there is a 5-point Likert Scale (1 meaning "not at all" and 5 meaning "very much") that needs to be answered.
Therapist's satisfaction of the use of VR as a tool for rehabilitation on ICU | Inclusion between 31/10/2022 and 31/10/2023. Screening for this particular outcome will happen during the 3-week-VR-training period for each patient.
  Motivation, time consuming, ... (through self-made questionnaire based on existing literature and approved by protocol). For every question there is a 5-point Likert Scale (1 meaning "not at all" and 5 meaning "very much") that needs to be answered.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Haghedooren, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
General data will be shared through a scientific article. No individual participant data will be shared.